CLINICAL TRIAL: NCT00588848
Title: Postoperative Management of Obstructive Sleep Apnea With CPAP vs. an Autoadjusting CPAP Device: a Randomized Controlled Single Center Trial
Brief Title: CPAP vs AutoCPAP for Treatment of Obstructive Sleep Apnea (OSA) in the Postoperative Setting
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with enrollment
Sponsor: MetroHealth Medical Center (Other)
Collaborators: ResMed (Industry); Great Lakes NeuroTechnologies Inc. (Industry)
Responsible Party: Principal Investigator, Dennis Auckley, MD, Associate Professor of Medicine, CWRU, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB07-00504
Record Dates: First submitted 2008-01-03; First posted 2008-01-09 (Estimated); Results first posted 2013-05-27 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea Hypopnea Syndrome; OSA; Postoperative; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autoadjusting CPAP (VPAP auto) (Experimental): The intervention will be the use of an Autoadjusting CPAP unit that will be applied to the subject during the 8 hours overnight the first night after surgery (study night). During this time, they will undergo a full night attended polysomnogram in their hospital room.
  Interventions: Device: Autoadjusting CPAP (VPAP Auto)
- CPAP arm (usual care) (Active Comparator): The intervention will be the use of the subject's own CPAP machine and this will be applied to the subject during the 8 hours overnight the first after surgery (study night). During the study night, they will undergo full polysomnography in their hospital room.
  Interventions: Device: CPAP

INTERVENTIONS:
Device: Autoadjusting CPAP (VPAP Auto) — An autoadjusting CPAP unit is used in place of subject's own CPAP unit during the night of the polysomnography study (the first night after surgery).
  Other Names: VPAP Auto
  Arms: Autoadjusting CPAP (VPAP auto)
Device: CPAP — Subject's own CPAP unit is applied to the subject during the polysomnography study night (the first night after surgery)
  Arms: CPAP arm (usual care)

SUMMARY:
The purpose of this study is to determine if an Autoadjusting CPAP machine is better than the regular CPAP machine in treatment of Obstructive Sleep Apnea in the postoperative setting.

DETAILED DESCRIPTION:
The purpose of this study is to determine if an Autoadjusting CPAP machine is better than the regular CPAP machine in treatment of Obstructive Sleep Apnea in the postoperative setting.

Patients with known Obstructive Sleep Apnea who are on CPAP therapy at home and undergo an elective surgery (meeting specified inclusion and exclusion criteria) will be randomized to either using Autoadjusting CPAP vs their usual CPAP at their prescribed settings the night after surgery. During that night, they will be monitored with full polysomnography in their hospital bed.

ELIGIBILITY:
Inclusion Criteria:

1. Known OSA patients well-controlled by CPAP (not hypoxemic i.e. Oxygen Saturation (SaO2) ≥ 89% and post-treatment Apnea Hypopnea (AHI) <10) and compliant ( > 3 hours per night) presenting for elective inpatient surgery to MetroHealth Medical Center
2. Elective extremity or lower abdominal surgery
3. Age >18 years

Exclusion Criteria:

1. Surgery that may cause hypoxemia from causes other than the effect on upper airway patency e.g. any thoracic surgery, upper abdominal surgery, head and neck surgery.
2. Surgery on the upper-airway.
3. Any condition that may interfere with application of CPAP mask e.g. trauma, surgery on the face, vomiting, naso-gastric intubation etc.
4. OSA treated with a device other than CPAP e.g. Bilevel positive pressure or V-Positive Airway Pressure
5. OSA needing very high levels of CPAP i.e. > 16 cms to achieve adequate control
6. OSA or other underlying cardiopulmonary conditions that require supplemental oxygen
7. Patients with decompensated congestive heart failure or advanced Chronic Obstructive Pulmonary Disease (COPD) (FEV1<35% of predicted)
8. Patients with neuromuscular impairment
9. Patients with central sleep apnea
10. Pregnant patients
11. Decisional impaired subjects who are not able to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Inderjeet S Brar, MD, Principal Investigator — MetroHealth Medical Center, Case Western Reserve University; Dennis Auckley, MD, Principal Investigator — MetroHealth Medical Center, Case Western Reserve University
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Young T, Peppard PE, Gottlieb DJ. Epidemiology of obstructive sleep apnea: a population health perspective. Am J Respir Crit Care Med. 2002 May 1;165(9):1217-39. doi: 10.1164/rccm.2109080. PMID 11991871
- [Background] Bailey PL, Pace NL, Ashburn MA, Moll JW, East KA, Stanley TH. Frequent hypoxemia and apnea after sedation with midazolam and fentanyl. Anesthesiology. 1990 Nov;73(5):826-30. doi: 10.1097/00000542-199011000-00005. PMID 2122773
- [Background] Ostermeier AM, Roizen MF, Hautkappe M, Klock PA, Klafta JM. Three sudden postoperative respiratory arrests associated with epidural opioids in patients with sleep apnea. Anesth Analg. 1997 Aug;85(2):452-60. doi: 10.1097/00000539-199708000-00037. No abstract available. PMID 9249130
- [Background] Gupta RM, Parvizi J, Hanssen AD, Gay PC. Postoperative complications in patients with obstructive sleep apnea syndrome undergoing hip or knee replacement: a case-control study. Mayo Clin Proc. 2001 Sep;76(9):897-905. doi: 10.4065/76.9.897. PMID 11560300
- [Background] Gross JB, Bachenberg KL, Benumof JL, Caplan RA, Connis RT, Cote CJ, Nickinovich DG, Prachand V, Ward DS, Weaver EM, Ydens L, Yu S; American Society of Anesthesiologists Task Force on Perioperative Management. Practice guidelines for the perioperative management of patients with obstructive sleep apnea: a report by the American Society of Anesthesiologists Task Force on Perioperative Management of patients with obstructive sleep apnea. Anesthesiology. 2006 May;104(5):1081-93; quiz 1117-8. doi: 10.1097/00000542-200605000-00026. No abstract available. PMID 16645462

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only 11 subjects were recruited but only 8 successfully completed the study (3 of the subjects randomized to the use of their usual CPAP slept less than 10 minutes on their night after surgery and thus were excluded from further analysis as the outcomes are based on events during sleep). This resulted in early termination of the study.
Pre-assignment Details: No significant events to report.
Groups:
- AUTOCPAP: An Autoadjusting CPAP unit will be applied to the subject during the 8 hours overnight the first night after surgery (study night)
  Autoadjusting Continuous Positive Airway Pressure (VPAP Auto) : An autoadjusting CPAP unit is used in place of subject's own CPAP unit during the night of the study (the first night after surgery).
- CPAP: Subject's own CPAP machine will be applied to the subject during the 8 hours overnight the first after surgery (study night)
  Continuous Positive Airway Pressure (CPAP) : Subject's own CPAP unit is applied to the subject during the study night (the first night after surgery)
Period: Overall Study
Arm/Group | AUTOCPAP | CPAP
Started | 3 | 8
Completed | 3 | 5
Not Completed | 0 | 3
Not completed — Physician Decision | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AUTOCPAP | CPAP | Total
Number analyzed (Participants) | 3 | 8 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 8 | 11
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (9.0) | 52.5 (7.5) | 51.2 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 8 | 11

OUTCOME MEASURES:

1. Primary Outcome: Sleep Related Hypoxemia
Time Frame: On postoperative night number 1 from 2200 to 0600. Study participation will end within 72 hours of admission.
Population: 3 of the subjects randomized to the use of their usual CPAP slept less than 10 minutes on their night after surgery and thus were excluded from further analysis as the outcomes are based on events during sleep.
Measure: Mean (Full Range); unit: Percentage of time < 90% saturation
Arm/Group | AUTOCPAP | CPAP
Number analyzed (Participants) | 3 | 5
Percentage of time < 90% saturation | 10.5 [0 to 52.0] | 7.1 [0 to 30.1]

2. Secondary Outcome: Apnea-Hypopnea Index (AHI)
Description: Events are defined as apneas and hypopneas. AHI values are typically categorized as 5-14.9 events/hr = mild; 15-29.9 events/hr = moderate; and >= 30 events/hr = severe
Time Frame: On postoperative night number 1 from 2200 to 0600. Study participation will end within 72 hours of admission.
Population: 3 of the subjects randomized to the use of their usual CPAP slept less than 10 minutes on their night after surgery and thus were excluded from further analysis as the outcomes are based on events during sleep. Study was terminated early due to enrollment problems.
Measure: Mean (Full Range); unit: events per hour
Arm/Group | AUTOCPAP | CPAP
Number analyzed (Participants) | 3 | 5
events per hour | 2.1 [0 to 5.5] | 1.2 [0 to 3.5]

3. Secondary Outcome: Cardiopulmonary Complications
Description: Predefined cardiopulmonary complications: Myocardial Infarction, Arrhythmia, new onset Heart Failure, Stroke
Time Frame: 72 hours
Population: None in either group
Measure: Count of Participants; unit: Participants
Arm/Group | Autoadjusting CPAP (VPAP Auto) | CPAP Arm (Usual Care)
Number analyzed (Participants) | 3 | 5
Participants | 0 | 0

ADVERSE EVENTS:
Description: Method for collection was to include chart review for prespecified adverse events.
  0 adverse events were recorded during the study.
Arm/Group | AUTOCPAP | CPAP
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/8
Other Adverse Events (participants affected / at risk) | 0/3 | 0/8

LIMITATIONS AND CAVEATS:
Trial limitations include:

1. Insufficient enrollment to adequately analyze data

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No